CLINICAL TRIAL: NCT05803460
Title: Explore the Effects of Virtual Reality Based Natural Environment Intervention Programs on Improving Attention, Emotion, and Cognitive Function of Older People
Brief Title: Explore the Effects of Virtual Reality Natural Environment of Older People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: YM111067E
Record Dates: First submitted 2023-03-13; First posted 2023-04-07 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2023-04

CONDITIONS: Older People
Keywords: Elders; Attention; Emotion; natural environment; virtual reality

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The data collection will be carried out by a researcher who is blind to the intervention allocation, according to standard research guideline.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Actual nature group: Actual experience of nature environment (Experimental): actual natural environment; participants in this group engage in 20 minutes of seated meditation in a natural park.
  Interventions: Behavioral: Experimental group: Actual nature group
- Virtual nature group: virtual reality experience of nature environment (Experimental): virtual reality experience of nature environment; Participants watched a 20-minute video of a virtual natural environment filmed by researchers.
  Interventions: Behavioral: Experimental group: Virtual nature group
- Actual urban group: actual experience of city (Active Comparator): actual experience of city; participants in the group engage in 20 minutes of seated meditation in a safe urban area.
  Interventions: Behavioral: Control group: Actual urban group

INTERVENTIONS:
Behavioral: Experimental group: Actual nature group — Participants will go to the park and sit still for 20 minutes.The natural environment site is the same as the video scenes used in the virtual natural environment intervention, located in a natural park in Taipei City.
  Arms: Actual nature group: Actual experience of nature environment
Behavioral: Experimental group: Virtual nature group — Participants will experience the virtual reality natural environment by the researcher for 20 minutes.The 360-degree panoramic natural environment scenes were from a natural park in Taipei City.Considering the elderly user experience, this study utilized standalone immersive virtual reality headset. Once wearing the goggles in a comfortable seated position, participants engaged in a 20-minute virtual reality environment experience.
  Arms: Virtual nature group: virtual reality experience of nature environment
Behavioral: Control group: Actual urban group — Participants will sit still for 20 minutes in a city environment.The urban environment is selected within the community's urban landscape.
  Arms: Actual urban group: actual experience of city

SUMMARY:
The objective of this study is to evaluate the effectiveness of virtual natural environment interventions on attention and mood among community-dwelling older adults in Taiwan. It was hypothesized that virtual reality combined with natural environments will improve attention to varying degrees and produce mood and physiological health outcomes in the elderly. This will be assessed by comparing the effects of virtual natural interventions with actual urban and natural interventions. Participants will randomly assign to virtual nature, actual nature, or actual urban group for a single 20-minute environmental session.

DETAILED DESCRIPTION:
This study will examine the effect of virtual natural environment intervention on attention and mood among community-dwelling older adults in Taiwan. This consist 3 parallel groups and 2 assessment periods. Participants in communities will be randomly assigned to virtual nature, actual nature, or actual urban group for a single 20-minute environmental session. Data will be collected at baseline and after intervention. This study recruits older adults from community locations in Taipei, Taiwan. Since no similar studies have been conducted before, the medium effect size 0. 25 is assumed, using the F-test analysis of variance, α = 0.05, power = 0.80, calculated the required total of 120 participants. Data is collected using mood and restorative questionnaires, attention tests, and a digital heart variability device. Statistical analyses will be performed using generalized estimating equations.

ELIGIBILITY:
Inclusion Criteria:

1. Age 65 years and older
2. Cognitive function is normal (SPMSQ >8)(The SPMSQ test was performed before the intervention to screen the cognitive function of the subjects).
3. The subjects can communicate in Chinese or Taiwanese.

Exclusion criteria:

1. Diseases affecting the results of the study, such as mental illness
2. Vision or hearing problems
3. Diseases transmitted by eyes or skin

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-04-07 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Digit span test | Baseline and 20 minutes
  To measure attention.
Trail Making Test | Baseline and 20 minutes
  To measure attention.
The Positive and Negative Affect Schedule | Baseline and 20 minutes
  To measure emotion.

SECONDARY OUTCOMES:
Blood pressure, heart rate and heart rate variability | Baseline and 20 minutes
  measure the participant's sitting blood pressure, heartbeat and heart rate variability.

OTHER OUTCOMES:
Perceived Restorativeness Scale | Baseline and 20 minutes
  To measure sleep status in the past month.

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Chen Chou, Ph.D, Principal Investigator — Nursing
Locations (1):
- National Yang Ming Chiao Tung University, Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No